CLINICAL TRIAL: NCT02765971
Title: The Efficacy of Chewing Gums Versus Laxatives in Early Return of Bowel Function After Cesarean Section
Brief Title: The Efficacy of Chewing Gums Versus Laxative in Early Return of Bowel Function After CS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed M Maged, MD (Other)
Responsible Party: Sponsor-Investigator, Ahmed M Maged, MD, Assistant professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 143
Record Dates: First submitted 2016-04-30; First posted 2016-05-09 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Intestinal Recovery After Cesarean Section
Keywords: chewing gums; laxatives; bowel function
MeSH Terms: interventions — Chewing Gum; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- chewing gum group (Active Comparator): 180 women will receive sugarless gum after their operating room discharge by 3 hours for at least half an hour at two hours interval
  Interventions: Other: gums
- laxatives group (Active Comparator): 180 women will receive laxatives after their operating room discharge by 3 hours
  Interventions: Drug: picolax drops
- control (Placebo Comparator): they will not receive neither gum nor oral fluids. They will be on intravenous fluid. starting oral fluids after hearing intestinal sounds
  Interventions: Drug: normal saline

INTERVENTIONS:
Other: gums — Group A, 180 women will receive sugarless gum after their operating room discharge by 3 hours for at least half an hour at two hours interval.
  Other Names: non sweet gums
  Arms: chewing gum group
Drug: picolax drops — Group B, 180 women will receive laxatives after their operating room discharge by 3 hours.
  Arms: laxatives group
Drug: normal saline — Group C received 500 cc of normal saline, Intravenous fluid
  Other Names: .9%saline infusion
  Arms: control

SUMMARY:
540 consented women for being enrolled in this clinical trial and candidates for elective cesarean section will be divided into 3 groups:

* Group A, 180 women will receive sugarless gum after their operating room discharge by 3 hours for at least half an hour at two hours interval.
* Group B, 180 women will receive laxatives after their operating room discharge by 3 hours.
* Group C, 180 women as control group, they will not receive neither gum nor oral fluids. They will be on intravenous fluid. starting oral fluids after hearing intestinal sounds .

DETAILED DESCRIPTION:
540 consented women for being enrolled in this clinical trial and candidates for elective cesarean section will be divided into 3 groups:

* Group A, 180 women will receive sugarless gum after their operating room discharge by 3 hours for at least half an hour at two hours interval.
* Group B, 180 women will receive laxatives after their operating room discharge by 3 hours.

Group C, 180 women as control group, they will not receive neither gum nor oral fluids. They will be on intravenous fluid. starting oral fluids after hearing intestinal sounds .

ELIGIBILITY:
Inclusion Criteria:

* all women undergoing elective cesarean section in Kasr Al AI Aini hospital will be candidate for this trial after full explanation of the trial and informed consent to be taken from the women.

Exclusion Criteria:

* cesarean hysterectomy,
* surgical management of severe postpartum hemorrhage
* previous bowel surgery
* women with history of drug consumption,especially opioids
* water and electrolyte disturbances
* pancreatitis or peritonitis
* inability to chew gum
* diabetes, pregnancies accompanied by coagulopathy like pre-eclampsia, hypothyroidism, muscular and neurological disorders
* postoperative admission to intensive care unit
* history of abdominal surgery except cesarean section
* history of postoperative ileus
* patients with drains

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 540 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
appearance of intestinal sounds postoperative evaluated by stethoscope | 4-6 hours after CS

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No